CLINICAL TRIAL: NCT02790359
Title: Carbon Dioxide Insufflation Versus Air Insufflation for Colonoscopy in Deeply Sedated Pediatric Patients: a Prospective, Randomized, Double Blind, Controlled Trial
Brief Title: Carbon Dioxide Insufflation Versus Conventional Air Insufflation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Diana Lerner, MD, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 728555
Record Dates: First submitted 2016-04-25; First posted 2016-06-03 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Abdominal Pain
Keywords: Carbon dioxide; Air; Colonoscopy
MeSH Terms: conditions — Abdominal Pain | interventions — Air; Carbon Dioxide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient group 1 (Active Comparator): Air
  Interventions: Other: Air
- Patient group 2 (Active Comparator): Carbon dioxide
  Interventions: Other: Carbon dioxide

INTERVENTIONS:
Other: Air — Group of patients who would receive air insufflation
  Arms: Patient group 1
Other: Carbon dioxide — Group of patients who would receive carbon dioxide insufflation
  Arms: Patient group 2

SUMMARY:
The safety and effectiveness of esophagogastroduodenoscopy and colonoscopy in the detection of gastrointestinal-tract pathology in children has been established during the last three decades. Insufflation of the intestinal tract, usually with room air, is necessary to improve visualization during the procedure; however, air in the bowels can also result in abdominal distension and increased pain. This potential discomfort associated with upper endoscopy and colonoscopy may be an important barrier to patients undergoing this procedure. Insufflation with carbon dioxide is another method used in endoscopic procedures for distention of the lumen and is currently used at the Children's Hospital of Wisconsin based on provider preference. The aim of this study is to perform a randomized controlled trial comparing insufflation with room air to carbon dioxide in patients undergoing routine upper endoscopy and colonoscopy. The investigators primary outcome is measurement of patient comfort level as measured by pain scores during recovery. The investigators hypothesize that carbon dioxide insufflation during endoscopy and colonoscopy improves patient comfort level as compared with insufflation with room air. Secondary outcome measures include changes in end tidal carbon dioxide, time to discharge, duration of colonoscopy and cecal intubation rate, changes in abdominal girth, rescue pain medications used during recovery and post-procedure events. This is a prospective randomized single-blinded study. The investigators will recruit consecutive patients, between the ages of 8 and 21 years, scheduled for elective outpatient upper endoscopy and colonoscopy at children's hospital of Wisconsin from March 2015 until we reach target population numbers. The investigators will exclude all inpatients, non-English speaking patients, children under 8 years of age, patients undergoing colonic manometry studies, and patients with hemodynamic instability, gastrointestinal bleeding, acute abdomen, previous colectomy, oxygen-dependent pulmonary disease and obstructive sleep apnea requiring the use of continuous positive airway pressure device. On the basis of a computer-generated randomization scheme in a 1:1 ratio, patients will be assigned to receive room air or carbon dioxide for insufflation during colonoscopy. Power calculation was done and determined that we will need to enroll 100 patients in each arm of the study. Informed consent will be obtained from all patients by the endoscopist or gastrointestinal fellow.

ELIGIBILITY:
Inclusion Criteria:

* ages of 8 and 21 years
* elective outpatient upper endoscopy and colonoscopy

Exclusion Criteria:

* inpatients
* non-English speaking patients
* children under 8 years of age
* patients undergoing colonic manometry studies
* patients with hemodynamic instability
* GI bleeding
* acute abdomen
* previous colectomy
* oxygen-dependent pulmonary disease and obstructive sleep apnea

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Abdominal pain based on visual analog scale | 72 hours
  Participants abdominal pain score will be assessed based on visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No